CLINICAL TRIAL: NCT05980936
Title: Screening for Obstructive Sleep Apnea in the General Medical Ward in Tertiary Care Centers in the Middle East
Brief Title: Screening for Obstructive Sleep Apnea in Medical Patients
Status: Withdrawn | Type: Observational
Why Stopped: no patients found
Sponsor: Jordan Collaborating Cardiology Group (Other)
Responsible Party: Sponsor
Other Study IDs: IH.OSAScrnng.2023/2
Record Dates: First submitted 2023-07-20; First posted 2023-08-08 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive sleep apnea; Symptomatology; Middle East
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Mass Screening

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Screening for obstructive sleep apnea — Patient will be interviewed and asked of there are symptoms of snoring, day somnolence, chocking or gasping during sleep

SUMMARY:
Obstructive sleep apnea (OSA) is highly prevalent in the general population and is associated with multiple adverse cardiovascular consequences.

Screening for OSA is recommended in those with typical symptoms, such as daytime sleepiness, loud snoring, or abrupt awakenings with gasping or choking. Patients admitted to the general medical wards with these symptoms will be evaluated for the possibility of having OSA.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is a disease that is highly prevalent in all communities and is associated with adverse cardiovascular events.

Screening for OSA is recommended in men and women who have the typical symptoms, including snoring, daytime sleepiness, or abrupt awakenings with choking or gasping.

OSA screening is also recommended for those with resistant hypertension, bradyarrhythmias, and atrial fibrillation.

Heart failure patients should also be screened for OSA. It is very important to increase the use of OSA screening especially in patients admitted to the medical floor in tertiary care hospitals. No study has evaluated this topic in the Middle East in the past.

ELIGIBILITY:
Inclusion Criteria:

* Willing to sign an informed consent
* Patient is admitted to the medical ward in a tertiary hospital

Exclusion Criteria:

* Patients known to have obstructive sleep apnea.
* Patients younger than 18 years of age

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients without known OSA who are admitted to the general medical ward will be Screened for signs and symptoms of OSA by answering the questions that have the statement :Do you have...?". The symptoms include snoring, day time somnolesce, sudden chocking or gasping during sleep..
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-10-15 (Actual); Primary Completion 2025-02-15 (Actual); Study Completion 2025-02-22 (Actual)

PRIMARY OUTCOMES:
Number of Participants who are found to have obstructive sleep apnea | From date of study enrollment until the date of first documented diagnosis of obstructive sleep apnea, assessed up to 4 weeks.
  Those who are found to have symptoms of OSA will be referred for further evaluation to get the final diagnosis of OSA

CONTACTS AND LOCATIONS:
Locations (2):
- Jordan (2):
  - Ayman Hammoudeh, Amman
  - Istishari Hospital, Amman